CLINICAL TRIAL: NCT03998735
Title: Nornicotine in Smokeless Tobacco as a Precursor for Carcinogen Exposure
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2019NTLS123; SPH-2019-23251 (Other: University of Minnesota); NCT02499198 (obsolete NCT alias)
Record Dates: First submitted 2019-06-24; First posted 2019-06-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Smokeless Tobacco
MeSH Terms: conditions — Tobacco Use | interventions — Tobacco, Smokeless

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1 (N=15) (Experimental): 160 µg/g herbal snuff, median level found in commercial moist snuff
  Interventions: Drug: Herbal Snuff (Smokeless Tobacco)
- Group 2 (N=15) (Experimental): 70 µg/g herbal snuff, lowest level found in commercial moist snuff (rounded)
  Interventions: Drug: Herbal Snuff (Smokeless Tobacco)
- Group 3 (N=15) (Experimental): 3.5 µg/g herbal snuff, 5% of the lowest level found in commercial moist snuff
  Interventions: Drug: Herbal Snuff (Smokeless Tobacco)
- Group 4(N=10) (Active Comparator): 0 µg/g herbal snuff, control group will use unmodified herbal snuff
  Interventions: Drug: Herbal Snuff (Smokeless Tobacco)

INTERVENTIONS:
Drug: Herbal Snuff (Smokeless Tobacco) — 4 levels of [D4]nornicotine in herbal snuff

SUMMARY:
Our goal in this study is to investigate the extent of endogenous nitrosation of nornicotine in smokeless tobacco users as a function of nornicotine content in smokeless products. This study will lead to an understanding of the endogenous formation of NNN from nornicotine in humans, and will also investigate the effect of the reduction of nornicotine content in smokeless tobacco on the extent of endogenous NNN formation. The knowledge gained in this study will lead to the development of recommendations for the regulation, or potentially elimination, of nornicotine in smokeless tobacco products in order to minimize exposure to NNN in the users of these products.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult smokeless tobacco users 18-65 years of age, using at least 3 tins of product per week for 6 months;
* Used the same brand for >80% of their smokeless tobacco use over the course of at least 6 months, and used this brand exclusively for at least two weeks prior to the eligibility screening;
* Not smoking or using any other nicotine or tobacco product in the past 2 weeks (expired CO < 6 ppm);
* Participants are in good physical health (no unstable medical condition) and good general oral health as determined by the licensed medical professional;
* Participants are in stable, good mental health (e.g. not currently, within the past 6 months, experiencing unstable or untreated psychiatric diagnosis, including substance abuse) as determined by the licensed medical professional;
* Participants who are not taking any medications that affect relevant metabolic enzymes;
* Women who are not pregnant or nursing or planning to become pregnant;
* Participants have provided written informed consent to participate in the study.

Exclusion Criteria:

* Significant immune system disorders, respiratory diseases, kidney or liver diseases or any other medical disorders that may affect biomarker data as determined by the licensed medical professional;
* Vital signs out of range as determined by the licensed medical professional (participants failing for vital signs will be allowed to re-screen once):
* Evident poor oral health (significant gum recession, dental caries, tooth loss) as determined by the general oral health status check;
* Excessive drinking (e.g., 5 or more drinks daily) or problems with drinking or drugs (e.g., self-report of binge drinking alcohol or treatment for drug or alcohol abuse within last 3 months); to be assessed by PI or licensed medical professional;
* Regular smoking or tobacco use (e.g., greater than once a week) other than oral smokeless tobacco products;
* Currently (within the past 2 weeks) using nicotine replacement or other tobacco cessation products (to minimize confounding effects of another product);

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2021-10-19 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
To investigate endogenous formation of NNN in smokeless tobacco users. | 2 Weeks
  Presence of urinary [pyridine-D4]NNN ([D4]NNN)
To investigate endogenous formation of NNN in smokeless tobacco users. | 2 Weeks
  Level of urinary [pyridine-D4]NNN ([D4]NNN) present

CONTACTS AND LOCATIONS:
Overall Officials: Irina Stepanov, PhD, Principal Investigator — University of Minnesota, Division of Environmental Health Sciences
Locations (1):
- Masonic Cancer Center, Minneapolis, Minnesota, United States